CLINICAL TRIAL: NCT04566796
Title: Effectiveness of Sugammadex on Muscle Relaxant Reversal in Preterm Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Mohamed Osman, assistant professor of anesthesia Alexandria university, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 234
Record Dates: First submitted 2020-09-16; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Sugammadex
Keywords: Sugammadex; preterm neonates
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: via the closed envelope method
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group N) (Active Comparator): patients in this group will receive 0.02 mg/kg atropine with neostigmine 0.05 mg/kg IV. to reverse the action of the neuromuscular blocker given.
  Interventions: Drug: Neostigmine
- (Group S) (Experimental): the patients will receive Sugammadex 2mg/kg IV. As the reversal agent
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — give 2 mg/ kg as muscle reversal drug in premature infants
  Arms: (Group S)
Drug: Neostigmine — give 0.02 mg/ kg atropine and 0.05 mg/kg neostigmine IV. as muscle reversal drug in premature infants
  Arms: (Group N)

SUMMARY:
The primary aim of the work is to compare the efficacy of Sugammadex and neostigmine in reversing rocuronium-induced muscle relaxation to reach complete recovery of neuromuscular block (TOF ratio≥ 0.9) in preterm neonates.

The secondary aim is to evaluate the safety of using Sugammadex in preterm neonates and to detect any complications that may occur in this age group.

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates
* scheduled for elective inguinal hernia repair

Exclusion Criteria:

* drug hypersensitivity
* patient is with any diseases affecting the neuromuscular junction
* Patients with family history of malignant hyperthermia

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of reversal | immediately after the surgery
  Reversal time which is defined as time in seconds from the start of administration of sugammadex or neostigmine to recovery of TOF ratio to 0.9
Evaluation of recovery | immediately after the surgery
  Time for modified Aldrete score to reach 10

SECONDARY OUTCOMES:
number of patients with Complications | immediately after the surgery
  any complication during recovery will be noted

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Elshafie, Principal Investigator — Alexandria University
Locations (1):
- Alexandria university, Alexandria, Egypt